CLINICAL TRIAL: NCT05937386
Title: An Open-Label, Fixed-Sequence, Drug-Drug Interaction Study in Healthy Participants to Evaluate the Effect of AGMB-129 on the Pharmacokinetics of Midazolam, a Sensitive Index Substrate of CYP3A4
Brief Title: Drug-Drug Interaction Study With AGMB-129 and Midazolam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agomab Spain S.L. (Industry)
Responsible Party: Sponsor
Organization: Agomab Therapeutics NV (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AGMB-129-C104
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): AGMB-129 and MDZ
  Interventions: Drug: AGMB-129; Drug: MDZ

INTERVENTIONS:
Drug: AGMB-129 — Oral capsule
Drug: MDZ — Pre-filled oral syringes

SUMMARY:
This is a single-center, open-label, fixed-sequence, Phase 1 study in healthy adult participants to evaluate the effect of AGMB-129 on the PK of a single dose of MDZ in healthy participants.

A total of 14 participants will be enrolled and will receive study intervention in a fixed-sequence scheme. All IP will be administered orally and in fed conditions.

The total duration of involvement for each participant, screening through follow-up, will be approximately 6 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, between 18 and 55 years old (extremes included) on the date of signing the ICF.
2. Body weight of at least 50.0 kg for men and 45.0 kg for women, and a body mass index (BMI) between 19.0 and 30.0 kg/m2 (extremes included) at screening.
3. Must be in good health based on medical history, physical examination, vital signs, and 12-lead ECG in the opinion of the investigator at screening.
4. Total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be ≤1.5x upper limit of normal (ULN) at screening. Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator. Note: Participants with diagnosed Gilbert's syndrome with total bilirubin >1.5 ULN are eligible for the study if AST and ALT are ≤1.5x ULN.

Key Exclusion Criteria:

1. Known hypersensitivity to AGMB-129 ingredients or history of a significant allergic reaction to AGMB-129 ingredients as determined by the investigator.
2. Positive serology for hepatitis B virus surface antigen (HBsAg) or anti-hepatitis C virus [HCV] antibodies at screening, or history of hepatitis from any cause except for hepatitis A that was resolved at least 3 months prior to the first IP administration.
3. History of or a current immunosuppressive condition, including positive human immunodeficiency virus types 1 or 2 (HIV-1 [2]) antibodies at screening.
4. Current or history of vasculitis, valvular heart disease, or large vessel vascular disease (such as aneurism or dissection) at screening.
5. Any illness, judged by the investigator as clinically significant, in the 3 months prior to the first IP administration.
6. Presence or sequelae of gastrointestinal, liver, kidney (estimated glomerular filtration rate [eGFR] ≤80 mL/min/1.73 m² using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs at screening.
7. History of malignancy within the past 5 years prior to screening, except for excised and curatively treated non-metastatic basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of cervix which is considered cured with minimal risk of recurrence.
8. History or presence of clinically significant abnormalities detected on 12-lead ECG of either rhythm or conduction, e.g., known long QT syndrome or a QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 ms detected on the 12-lead ECG at screening or Day 1 predose. A first-degree atrioventricular block will not be considered as a clinically significant abnormality.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Cmax for MDZ | Day 1 to Day 13
Cmax for 1-OH-midazolam | Day 1 to Day 13
AUC0-∞ for MDZ | Day 1 to Day 13
AUC0-∞ for 1-OH-midazolam | Day 1 to Day 13

SECONDARY OUTCOMES:
Cmax for AGMB-129 | Day 3 to Day 14
Cmax for MET-154 | Day 3 to Day 14
Cmax for MET-158 | Day 3 to Day 14
AUC0-t for AGMB-129 | Day 3 to Day 14
AUC0-t for MET-154 | Day 3 to Day 14
AUC0-t for MET-158 | Day 3 to Day 14
AUC0-24 for AGMB-129 | Day 3 to Day 14
AUC0-24 for MET-154 | Day 3 to Day 14
AUC0-24 for MET-158 | Day 3 to Day 14
Number of participants with adverse events | From Screening to Day 15
  To evaluate the safety and tolerability of AGMB-129 in terms of adverse events at every visit
Number of participants with abnormal clinical laboratory values | From Screening to Day 15
  To evaluate the safety and tolerability of AGMB-129 in terms of abnormal laboratory parameters at every visit
Number of participants with abnormal vital signs | From Screening to Day 15
  To evaluate the safety and tolerability of AGMB-129 in terms of vital signs at every visit
Number of participants with abnormal physical exams | From Screening to Day 15
  To evaluate the safety and tolerability of AGMB-129 in terms of physical exams at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Wiesel, MD, Study Director — Agomab Therapeutics
Locations (1):
- SGS Belgium, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No